CLINICAL TRIAL: NCT04404790
Title: Phase I Clinical Trial of the Tolerance and Pharmacokinetics of Anfibatide in Health Volunteer
Brief Title: Antiplatelet Thrombolysin (Anfibatide) Phase 1 Clinical Trial in Healthy Volunteers
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Optimization of protocol
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZK-APT-201803
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Antiplatelet Drug
MeSH Terms: interventions — agkisacucetin protein, Agkistrodon acutus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Anfibatide 5 IU/60kg (Experimental): Ten subjects will injected with the dose of 5 IU/60kg of Anfibatide with 5 minutes.
  Interventions: Drug: Anfibatide 5 IU/60kg
- Anfibatide 5 IU/60kg+0.002 IU/kg/h (Experimental): Four or fourteen subjects will injected with the dose of 5 IU/60kg of Anfibatide with 5 minutes follow by the dose of 0.002 IU/kg/h continuous intravenous infusion with 48 hours.
  Interventions: Drug: Anfibatide 5 IU/60kg +0.002 IU/kg/h
- Anfibatide 5 IU/60kg+0.004 IU/kg/h (Experimental): Four or fourteen subjects will injected with the dose of 5 IU/60kg of Anfibatide with 5 minutes follow by the dose of 0.004 IU/kg/h continuous intravenous infusion with 48 hours.
  Interventions: Drug: Anfibatide 5 IU/60kg +0.004 IU/kg/h
- Anfibatide 5 IU/60kg+0.008 IU/kg/h (Experimental): Four or fourteen subjects will injected with the dose of 5 IU/60kg of Anfibatide with 5 minutes follow by the dose of 0.008 IU/kg/h continuous intravenous infusion with 48 hours.
  Interventions: Drug: Anfibatide 5 IU/60kg +0.008 IU/kg/h
- Anfibatide 7 IU/60kg (Experimental): Ten subjects will injected with the dose of 7 IU/60kg of Anfibatide with 5 minutes.
  Interventions: Drug: Anfibatide 7 IU/60kg
- Anfibatide 7 IU/60kg+0.002 IU/kg/h (Experimental): Four or fourteen subjects will injected with the dose of 7 IU/60kg of Anfibatide with 5 minutes follow by the dose of 0.002 IU/kg/h continuous intravenous infusion with 48 hours.
  Interventions: Drug: Anfibatide 7 IU/60kg +0.002 IU/kg/h
- Anfibatide 7 IU/60kg+0.004 IU/kg/h (Experimental): Four or fourteen subjects will injected with the dose of 7 IU/60kg of Anfibatide with 5 minutes follow by the dose of 0.004 IU/kg/h continuous intravenous infusion with 48 hours.
  Interventions: Drug: Anfibatide 7 IU/60kg +0.004 IU/kg/h
- Anfibatide 7 IU/60kg+0.008 IU/kg/h (Experimental): Four or fourteen subjects will injected with the dose of 7 IU/60kg of Anfibatide with 5 minutes follow by the dose of 0.008 IU/kg/h continuous intravenous infusion with 48 hours.
  Interventions: Drug: Anfibatide 7 IU/60kg +0.008 IU/kg/h

INTERVENTIONS:
Drug: Anfibatide 5 IU/60kg — 5 IU/60kg IV administration of Anfibatide with 5 minutes
  Arms: Anfibatide 5 IU/60kg
Drug: Anfibatide 5 IU/60kg +0.002 IU/kg/h — 5 IU/60kg IV administration of Anfibatide with 5 minutes follow by the dose of 0.002 IU/kg/h continuous intravenous infusion with 48 hours
  Arms: Anfibatide 5 IU/60kg+0.002 IU/kg/h
Drug: Anfibatide 5 IU/60kg +0.004 IU/kg/h — 5 IU/60kg IV administration of Anfibatide with 5 minutes follow by the dose of 0.004 IU/kg/h continuous intravenous infusion with 48 hours
  Arms: Anfibatide 5 IU/60kg+0.004 IU/kg/h
Drug: Anfibatide 5 IU/60kg +0.008 IU/kg/h — 5 IU/60kg IV administration of Anfibatide with 5 minutes follow by the dose of 0.008 IU/kg/h continuous intravenous infusion with 48 hours
  Arms: Anfibatide 5 IU/60kg+0.008 IU/kg/h
Drug: Anfibatide 7 IU/60kg — 7 IU/60kg IV administration of Anfibatide with 5 minutes
  Arms: Anfibatide 7 IU/60kg
Drug: Anfibatide 7 IU/60kg +0.002 IU/kg/h — 7 IU/60kg IV administration of Anfibatide with 5 minutes follow by the dose of 0.002 IU/kg/h continuous intravenous infusion with 48 hours
  Arms: Anfibatide 7 IU/60kg+0.002 IU/kg/h
Drug: Anfibatide 7 IU/60kg +0.004 IU/kg/h — 7 IU/60kg IV administration of Anfibatide with 5 minutes follow by the dose of 0.004 IU/kg/h continuous intravenous infusion with 48 hours
  Arms: Anfibatide 7 IU/60kg+0.004 IU/kg/h
Drug: Anfibatide 7 IU/60kg +0.008 IU/kg/h — 7 IU/60kg IV administration of Anfibatide with 5 minutes follow by the dose of 0.008 IU/kg/h continuous intravenous infusion with 48 hours
  Arms: Anfibatide 7 IU/60kg+0.008 IU/kg/h

SUMMARY:
This is a phase 1, dose-escalation, and multidose study, aiming to investigate the tolerability, safety and pharmacokinetics of Anfibatate in healthy subjects. The study is divided into 2 intravenous single groups and 3 continuous administration groups. The dose of Anfibatate from 5 IU/60kg to 7 IU/60kg in intravenous single groups. The dose of Anfibatate from 0.002 IU/kg/h, 0.004 IU/kg/h to 0.008 IU/kg/h in continuous administration groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy subjects between the ages of 18 to 40 years（including）.
2. The body mass index（BMI）， in the range of 19 ~ 24 (including).
3. Medical history without heart, liver, kidney, digestive tract, nervous system, metabolic, ulcer, obvious bleeding, and history of drug allergy or postural hypotension.
4. According to the medical history, physical examination, vital signs, chest radiograph, 12-lead ECG, coagulation routine, stool routine and occult blood test, as well as the laboratory results of blood and urine, the subjects are healthy.
5. The subjects do not take any medicine in the past two weeks.
6. Willingness to participate the study and sign the written Informed Consent Form.
7. Non-lactating women willingness to use adequate contraceptive measures (including abstinence, intrauterine device, diaphragm and spermicide) during the study (screening period to 1 week after administration). Men are willing to use approved methods of contraception (including condoms and spermicides or oral, implanted or injectable contraceptives by their partners, intrauterine device, diaphragms and spermicides). Subjects do not plan to donate sperm or eggs within two weeks after drug administration.

Exclusion Criteria:

1. Abnormal with the safety evaluation is considered to be clinical significance in screening period as judged by the researcher.
2. Subjects with history of hepatitis B virus, hepatitis C virus, human immunodeficiency virus and syphilis virus infection;
3. Excessive smoking (>5 cigarettes/day) or do not interrupt smoke during the study.
4. Intake of more than 25g of alcohol per day (equivalent to 750 mL of beer or 250 mL of wine, or 75 mL of white wine of 38 °, or 50 mL of white wine of ≥40 ° ). Subject who are positive for alcohol breath test or cannot stop drinking during the study.
5. Women with pregnant, lactating or menstruating.
6. History of previous hemoptysis, blood stool, skin mucosal bleeding points, etc., or bleeding tendency (patients with gingival, nasal, skin, mucosal bleeding, hemoptysis).
7. History of active bleeding (peptic ulcer, hemorrhoids, active tuberculosis, subacute bacterial endocarditis, etc.).
8. The examination show arteriovenous malformation, hemangioma and other vascular abnormalities.
9. The examination show that there is hemorrhage in the fundus.
10. The platelet count is less than 150×109/L.
11. History of trauma (craniocerebral trauma, etc.) within 1 year.
12. History of unexplained syncope or convulsions.
13. History of autoimmune diseases, such as systemic lupus erythematosus.
14. History of organic or mental illnesses or disabilities.
15. According to the judgment by the researchers, subjects with low possibility of enrollment (such as weak body, etc.).
16. Donation of blood in the last 3 months or participation in other clinical trials in the last 3 months.
17. Previously recruited into other clinical studies of the product.
18. Mental, psychological, or language disorders that prevent understanding or cooperation.
19. Unwilling or unable to comply with the study schedule or procedure.
20. Unfit to participate in the study for any other reason.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Bleeding events | 7 days after drug administration
  Bleeding events are judged according to Bleeding Academic Research Consortium Definition for Bleeding criteria.

SECONDARY OUTCOMES:
Cmax | 7 days after drug administration
  Peak concentration
Tmax | 7 days after drug administration
  Peak time
AUC(0-t) | 7 days after drug administration
  Area under curve 0-t
AUC(0-∞) | 7 days after drug administration
  Area under curve 0-∞
T1/2 | 7 days after drug administration
  Half life
Inhibition of platelet aggregation | 7 days after drug administration
  Inhibition rate of platelet aggregation is measured by chrono-log700.
corrected QT interval | 7 days after drug administration
  Corrected QT interval is measured by 12-lead ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Ningru Zhang, Study Director — Bengbu Medical College First Hospital
Locations (1):
- Bengbu Medical College First Hospital, Bengbu, Anhui, China